CLINICAL TRIAL: NCT00148369
Title: A Multi-Center, Observational Safety Registry of Subjects With Idiopathic Parkinson's Disease Previously Treated With Intraputaminal Infusion of Liatermin
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Other Study IDs: 20040256
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2010-02-19 (Estimated); Status verified 2010-02

CONDITIONS: Idiopathic Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: None Retained — none collected.

GROUPS / COHORTS (1):
- Observational Group: Subjects previously administered GDNF and have discontinued the drug.
  Interventions: Drug: Safety observation

INTERVENTIONS:
Drug: Safety observation — Subjects previously enrolled in a GDNF protocol observed for 2 years after discontinuation of drug.

SUMMARY:
The primary purpose of this study is to evaluate clinical and serologic outcomes after the discontinuation of liatermin therapy as assessed by development of new clinical conditions beyond those expected in patients with advancing Parkinson's disease. In addition, the development or resolution of anti-r-metHuGDNF binding and neutralizing antibodies will be monitored.

ELIGIBILITY:
Inclusion Criteria: - Subjects must have a diagnosis of bilateral, idiopathic Parkinson's Disease who have been enrolled and treated with intraputaminal infusion of liatermin in a previous Amgen/Medtronic-sponsored trial (protocols 20010109 or 20030160) or the Bristol open-label study - At time of implant (Study 20030168), subjects need to have been 35 to 70 years of age

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with idiopathic Parkinson's Disease
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2005-06; Primary Completion 2006-11 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com